CLINICAL TRIAL: NCT00705419
Title: COVER - Continuing Observation After Vicriviroc (VCV) Exposure Registry
Brief Title: Registry to Assess Long-term Outcome in HIV Subjects Who Participated in Phase 2 and 3 Clinical Trials Involving Vicriviroc (Study P04999)
Acronym: COVER
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04999
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Previous vicriviroc 30 mg QD: Subjects who previously received vicriviroc 30 mg daily in a Phase 2 or 3 clinical trial.
  Interventions: Drug: Vicriviroc maleate
- Previous vicriviroc 20 mg QD: Subjects who previously received vicriviroc 20 mg daily in a Phase 2 or 3 clinical trial.
  Interventions: Drug: Vicriviroc maleate
- Control Group: Subjects who previously received active control or placebo in a Phase 2 or 3 clinical trial involving vicriviroc.
  Interventions: Drug: Placebo; Drug: Emtricitabine 200 mg/ tenofovir disoproxil fumarate 300 mg

INTERVENTIONS:
Drug: Vicriviroc maleate — Follow-up for subjects who previously received 30 mg tablet administered once daily according to the parent protocol.
  Other Names: SCH 417690
  Groups: Previous vicriviroc 30 mg QD
Drug: Vicriviroc maleate — Follow-up for subjects who previously received 20 mg tablet administered once daily according to the parent protocol.
  Other Names: SCH 417690
  Groups: Previous vicriviroc 20 mg QD
Drug: Placebo — Follow-up for subjects who previously received placebo tablet administered once daily according to the parent protocol.
  Groups: Control Group
Drug: Emtricitabine 200 mg/ tenofovir disoproxil fumarate 300 mg — Follow-up for subjects who previously received active control consisting of emtricitabine 200 mg/ tenofovir disoproxil fumarate 300 mg combination tablet administered once daily according to the parent protocol.
  Other Names: Truvada
  Groups: Control Group

SUMMARY:
Nonrandomized, prospective, observational, multi-site registry to assess long-term safety, clinical outcome, deaths, and evolution of viral tropism in HIV subjects who completed or discontinued participation in Phase 2 or 3 clinical trials involving vicriviroc. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
A non-probability sampling method will be used. Subjects will be requested to enroll in the registry after having completed or discontinued participation in a Phase 2 or 3 study involving vicriviroc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have participated in a Phase 2 or 3 study involving vicriviroc, and must have received, but are no longer receiving study medication.

Exclusion Criteria:

* Unwillingness to participate in the registry or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will enroll subjects who received vicriviroc or control in a Phase 2 or 3 clinical trial (with the exception of P03802 and ACTG A5211 [and its rollover P04100]), and are no longer receiving study medication.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of malignancies, AIDS-defining events, other clinical events of importance, and death. | Information regarding clinical outcome will be collected every 6 months. Deaths will be collected on an ongoing basis.

SECONDARY OUTCOMES:
Incidence of change in plasma viral tropism, time to change in plasma viral tropism, and change in HIV RNA and CD4+ counts, if available. | Every 6 months.